CLINICAL TRIAL: NCT01741792
Title: An Open Label, Multicenter, Exploratory Phase 2 Study to Evaluate the Efficacy and Safety of the Bispecific T-Cell Engager (BiTE®) Blinatumomab in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Clinical Study With Blinatumomab in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT103-208; 2011-005781-38 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-12-05 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Relapsed DLBCL; Refractory DLBCL; adult DLBCL; Lymphoma; Non-Hodgkin Lymphoma; Lymphatic diseases; Lymphoproliferative disorders; bispecific antibody; anti-CD19; Immunotherapeutic treatment; Immunoproliferative disorders
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, Non-Hodgkin; Lymphatic Diseases; Lymphoproliferative Disorders; Immunoproliferative Disorders | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blinatumomab (Experimental): By study design, two dose regimens were assessed in this study. In Stage 1, Cohort 1, participants received blinatumomab in a dose-escalating manner: 9 µg/day for the first week, followed by 28 µg/day for the second week, then 112 µg/day for the remaining 6 weeks of treatment during cycle 1. In Cohort 2, the next participants enrolled and received a constant dose of 112 µg/day blinatumomab. The dosing regimen with the more favorable benefit-risk profile was then selected for Stage 2, Cohort 3.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Administered by continuous intravenous infusion over 8 weeks in the first cycle and 4 weeks in the second cycle.
  Other Names: AMG103; MT103; BLINCYTO®

SUMMARY:
The purpose of this study is to confirm whether the bispecific T-cell engager blinatumomab is effective and safe in the treatment of patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
DLBCL is an aggressive malignant disease which evolves from B-cells and affects mainly the lymphatic tissue. Due to its aggressive nature the disease is characterized by a fast course which is lethal without therapy. Potentially curative therapy options are available even at advanced stages. Standard-first line leads to a high initial response rate (85-90%) and an approximate cure rate of 50% of patients. Patients refractory to or with early relapse after this treatment (10-15%) have a very poor prognosis.

Blinatumomab is a bispecific single-chain antibody derivative against CD19 and CD3, designed to link B-cells and T-cells resulting in T-cell activation and a cytotoxic T-cell response against CD19 expressing cells.

This study consisted of a screening period, treatment period, and a follow-up efficacy and survival period. The core study comprises the treatment period to the 30 days after the last infusion. The first cycle consisted of a continuous intravenous (CIV) infusion over 8 weeks. Participants who achieved a Complete Response (CR) or Partial Response (PR) or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval. After the last treatment cycle, efficacy and survival follow-up visits occurred for up to 24 months from treatment start. Participants who relapsed during the follow-up period may have received an additional 8 weeks of treatment.

Two dose regimens were assessed in this study. Stage 1 comprised 2 dose cohorts. In Cohort 1, the first 6 participants were to receive blinatumomab in a dose-escalating manner: 9 µg/day for the first week, followed by 28 µg/day for the second week, then 112 µg/day for the remaining 6 weeks of treatment during Cycle 1. In Cohort 2, the next 6 participants enrolled were to receive a constant dose of 112 µg/day blinatumomab. Before the initiation of stage 2, a pre-planned data monitoring committee (DMC) meeting was held to assess the safety profile of Cohort 1 and Cohort 2. The dosing regimen with the more favorable benefit-risk profile was to be selected for Cohort 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diffuse Large B-Cell Lymphoma (DLBCL) who are refractory to first or later treatment or have a first relapse or later relapse not eligible for autologous hematopoietic stem cell transplant (HSCT) or relapsed post- autologous-HSCT
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Age ≥ 18 years
* Life expectancy of ≥ 12 weeks
* Cerebrospinal fluid (CSF) free of infiltration by DLBCL

Exclusion Criteria:

* History or presence of clinically relevant central nervous system (CNS) pathology as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis
* Current infiltration of CSF by DLBCL
* History of autoimmune disease with potential CNS involvement or current autoimmune disease
* Autologous HSCT within six weeks prior to start of blinatumomab treatment
* Prior allogeneic HSCT
* Cancer chemotherapy within two weeks prior to start of blinatumomab treatment
* Radiotherapy within four weeks prior to start of blinatumomab treatment
* Immunotherapy (e.g., rituximab) within four weeks prior to start of blinatumomab treatment
* Any investigational anti-lymphoma product within four weeks prior to start of blinatumomab treatment
* Treatment with any other investigational product after signature of informed consent
* Known hypersensitivity to immunoglobulins or to any other component of the study drug formulation
* Abnormal laboratory values indicative of inadequate renal or liver function
* History of malignancy other than non-Hodgkin's lymphoma (NHL) within five years prior to start of blinatumomab treatment with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix
* Active uncontrolled infection, any other concurrent disease or medical condition that is deemed to interfere with the conduct of the study as judged by the investigator
* Infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus or hepatitis C virus
* Pregnant or nursing women
* Previous treatment with blinatumomab
* Presence of human anti-murine antibodies (HAMA) at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: - MD, Study Director — Amgen
Locations (6):
- Germany (6):
  - Universitätsmedizin, Göttingen
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Schleswig Holstein, Kiel
  - Klinikum der Johannes-Gutenberg Universität, Mainz
  - Universitätsklinikum, Ulm
  - Universititätsklinikum, Würzburg

REFERENCES:
- [Derived] Zhu M, Wu B, Brandl C, Johnson J, Wolf A, Chow A, Doshi S. Blinatumomab, a Bispecific T-cell Engager (BiTE((R))) for CD-19 Targeted Cancer Immunotherapy: Clinical Pharmacology and Its Implications. Clin Pharmacokinet. 2016 Oct;55(10):1271-1288. doi: 10.1007/s40262-016-0405-4. PMID 27209293
- [Derived] Viardot A, Goebeler ME, Hess G, Neumann S, Pfreundschuh M, Adrian N, Zettl F, Libicher M, Sayehli C, Stieglmaier J, Zhang A, Nagorsen D, Bargou RC. Phase 2 study of the bispecific T-cell engager (BiTE) antibody blinatumomab in relapsed/refractory diffuse large B-cell lymphoma. Blood. 2016 Mar 17;127(11):1410-6. doi: 10.1182/blood-2015-06-651380. Epub 2016 Jan 11. PMID 26755709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with a diagnosis of diffuse large B-cell lymphoma (DLBCL) which was refractory to first or subsequent treatment or who had a first or later relapse and were not eligible for autologous hematopoietic stem cell transplant (HSCT), or relapsed after autologous HSCT were eligible to enrol.
  The primary analysis cut-off date was 10 July 2014.
Pre-assignment Details: The study was conducted sequentially in 2 stages and 3 cohorts: In Stage 1, Cohort 1 received an escalating dose of 9/28/112 µg/day blinatumomab and Cohort 2 received a constant dose of 112 µg/day for 8 weeks. In Stage 2, the Cohort 3 dose regimen was determined from the outcome of Cohorts 1 and 2.
Groups:
- Cohort 1: Blinatumomab 9/28/112 µg/d: Participants received blinatumomab administered via a continuous intravenous infusion (CIV) 9 µg/day for the first week, followed by 28 µg/day for the second week, then 112 µg/day for the remaining 6 weeks of treatment during Cycle 1. Participants who achieved a complete response (CR) or partial response (PR), or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
- Cohort 2: Blinatumomab 112 µg/d: Participants received blinatumomab administered CIV at a constant dose of 112 µg/day for 8 weeks of treatment during Cycle 1. Participants who achieved a CR or PR, or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
- Cohort 3: Blinatumomab 9/28/112 µg/d: Participants received blinatumomab administered CIV 9 µg/day for the first week, followed by 28 µg/day for the second week, then 112 µg/day for the remaining 6 weeks of treatment during Cycle 1. Participants who achieved CR or PR, or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
Period: Overall Study
Arm/Group | Cohort 1: Blinatumomab 9/28/112 µg/d | Cohort 2: Blinatumomab 112 µg/d | Cohort 3: Blinatumomab 9/28/112 µg/d
Started | 9 (3 participants were not considered evaluable and were replaced as specified in the protocol.) | 2 (Cohort 2 was closed to enrollment on recommendation of the data monitoring committee) | 14
Efficacy Set | 7 (Completed > 7 days of infusion on the highest intended dose level or discontinued due to progression) | 1 (Completed > 7 days of infusion on the highest intended dose level or discontinued due to progression) | 13 (Completed > 7 days of infusion on the highest intended dose level or discontinued due to progression)
Completed | 3 | 1 | 2
Not Completed | 6 | 1 | 12
Not completed — Death | 6 | 1 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Blinatumomab 9/28/112 µg/d | Cohort 2: Blinatumomab 112 µg/d | Cohort 3: Blinatumomab 9/28/112 µg/d | Total
Number analyzed (Participants) | 9 | 2 | 14 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (7.8) | 64.5 (13.4) | 57.1 (13.6) | 62.9 (13.3)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 0 | 4 | 11
  Male | 2 | 2 | 10 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  White | 9 | 2 | 14 | 25
Relapsed/refractory Status to Last Prior Treatment [Number; unit: participants]
  Relapsed | 4 | 1 | 4 | 9
  Refractory | 5 | 1 | 10 | 16
Number of Previous Autologous Hematopoietic Stem Cell Transplants (HSCT) [Number; unit: participants]
  None | 7 | 1 | 10 | 18
  ≥ 1 | 2 | 1 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate During Treatment Cycle 1
Description: Overall response within the first treatment cycle was assessed according to Cheson criteria by a central reader. Response was evaluated using computerized tomography (CT) scans and positron emission tomography (PET) (to assess nodal disease/organ enlargement due to nodal/diffuse infiltration), and bone marrow biopsy (to assess bone marrow infiltration). Overall objective response rate (ORR) is the percentage of participants with a best overall response of complete response (CR) or partial response (PR).
  Complete response is defined as the disappearance of all evidence of disease and partial response is defined as regression of measureable disease and no new sites.
Time Frame: During the first 8 weeks
Population: Efficacy Set includes all participants who completed at least 7 days of infusion on the highest intended dose level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1: Blinatumomab 9/28/112 μg/d: Participants received blinatumomab administered via a continuous intravenous infusion (CIV) 9 µg/day for the first week, followed by 28 µg/day for the second week, then 112 µg/day for the remaining 6 weeks of treatment during Cycle 1. Participants who achieved a complete response (CR) or partial response (PR), or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
- Cohort 2: Blinatumomab 112 μg/d: Participants received blinatumomab CIV at a constant dose of 112 µg/day for 8 weeks of treatment during Cycle 1. Participants who achieved a CR or PR, or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
- Cohort 3: Blinatumomab 9/28/112 μg/d: Participants received blinatumomab administered CIV 9 µg/day for the first week, followed by 28 µg/day for the second week, then 112 µg/day for the remaining 6 weeks of treatment during Cycle 1. Participants who achieved CR or PR, or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 7 | 1 | 13
percentage of participants | 57.1 [18.4 to 90.1] | 100.0 [2.5 to 100.0] | 30.8 [9.1 to 61.4]

2. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response
Description: Response within the first treatment cycle was assessed according to Cheson criteria by a central reader. Response was evaluated using computerized tomography (CT) scans and positron emission tomography (PET) (to assess nodal disease/organ enlargement due to nodal/diffuse infiltration), and bone marrow biopsy (to assess bone marrow infiltration). Complete response is defined as the disappearance of all evidence of disease.
Time Frame: During the first 8 weeks
Population: Efficacy set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 7 | 1 | 13
percentage of participants | 28.6 [3.7 to 71.0] | 0 [0.0 to 97.5] | 15.4 [1.9 to 45.4]

3. Secondary Outcome: Percentage of Participants With a Best Overall Response of Partial Response
Description: Response within the first treatment cycle was assessed according to Cheson criteria by a central reader. Response was evaluated using computerized tomography (CT) scans and positron emission tomography (PET) (to assess nodal disease/organ enlargement due to nodal/diffuse infiltration), and bone marrow biopsy (to assess bone marrow infiltration). Partial response is defined as regression (<50% decrease in size of masses) of measureable disease and no new sites.
Time Frame: During the first 8 weeks
Population: Efficacy set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 7 | 1 | 13
percentage of participants | 28.6 [3.7 to 71.0] | 100.0 [2.5 to 100.0] | 15.4 [1.9 to 45.4]

4. Secondary Outcome: Duration of Objective Response
Description: The time from documentation of the first assessment of either partial or complete response until the start of new anti-tumor treatment (excluding any stem cell transplantation), progression of disease, or death, whichever is the earliest event. A patient who did not have new anti-tumor treatment (excluding any stem cell transplantation), progression of disease, or death was censored at last tumor assessment date. Disease progression is defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: From first infusion of blinatumomab until the end of study; median follow-up time for duration of response was 23.7 months.
Population: Efficacy set with an overall objective response of CR or PR during the first treatment cycle
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 4 | 1 | 4
months | 8.7 [0.9 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | 4.0 [1.9 to NA] — Could not be estimated due to the low number of events

5. Secondary Outcome: Duration of Complete Response
Description: The time from documentation of the first assessment of complete response until the start of new anti-tumor treatment (excluding any stem cell transplantation), progression of disease, or death, whichever is the earliest event. A patient who did not have new anti-tumor treatment (excluding any stem cell transplantation), progression of disease, or death was censored at last tumor assessment date. Disease progression is defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: as for outcome 4
Population: Efficacy set with a best overall response of CR during the first treatment cycle
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 2 | 0 | 2
months | NA [11.6 to NA] — Could not be estimated due to the low number of events |  | NA [5.9 to NA] — Could not be estimated due to the low number of events

6. Secondary Outcome: Duration of Partial Response
Description: The time from documentation of the first assessment of partial response until the start of new anti-tumor treatment (excluding any stem cell transplantation), progression of disease, or death, whichever is the earliest event. A patient who did not have new anti-tumor treatment (excluding any stem cell transplantation), progression of disease, or death was censored at last tumor assessment date. Disease progression is defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: as for outcome 4
Population: Efficacy set with a best overall response of PR during the first treatment cycle
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 2 | 1 | 2
months | 3.3 [0.9 to 5.8] | NA [NA to NA] — Could not be estimated due to the low number of events | 2.0 [1.9 to 2.1]

7. Secondary Outcome: Progression-free Survival (PFS)
Description: The time from the date of first blinatumomab infusion until the date of diagnosis of progression of lymphoma, the start date of new anti-tumor treatment (excluding any stem cell transplantation) or date of death, whichever is the earliest. Patients alive who did not have progression or new anti-tumor treatment (excluding any stem cell transplantation) were censored at last date of tumor assessment.
Time Frame: From first infusion of blinatumomab until the end of study; median time on follow-up for PFS was 27.0 months.
Population: Efficacy set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 7 | 1 | 13
months | 3.7 [0.7 to 14.1] | NA [NA to NA] — Could not be estimated due to the low number of events | 1.6 [0.6 to 4.6]

8. Secondary Outcome: Overall Survival (OS)
Description: The time from the date of first blinatumomab infusion until death as a result of any cause. Patients still alive were censored on the last documented visit date or the date of the last phone contact when the patient was last known to have been alive. For patients who withdrew their informed consent, only information until the date of withdrawal was analyzed.
Time Frame: From the first infusion of blinatumomab until the end of study; median time on follow-up for overall survival was 26.6 months.
Population: Efficacy set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 7 | 1 | 13
months | 20.1 [2.3 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | 3.6 [1.5 to 14.8]

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events were evaluated for severity according to the grading scale provided in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.0.
  An adverse event or suspected adverse drug reaction was considered "serious" if it resulted in one of the following outcomes:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant incapacity or substantial disruption to conduct normal life functions;
  * Was a congenital anomaly or birth defect;
  * Was a medically important condition.
  The Investigator used medical judgment to determine whether there was a causal relationship (ie, related [reasonably possible] or unrelated [not reasonably possible]) between an adverse event and blinatumomab.
Time Frame: From the first dose of blinatumomab until up to 30 days after the last dose or until the data cut-off date of 10 July 2014, whichever occurred first; the overall median duration of treatment exposure was 46.8 days.
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Cohort 1: Blinatumomab 9/28/112 μg/d | Cohort 2: Blinatumomab 112 μg/d | Cohort 3: Blinatumomab 9/28/112 μg/d
Number analyzed (Participants) | 9 | 2 | 14
participants
  Any adverse event (AE) | 9 | 2 | 14
  AE of Grade ≥ 3 | 9 | 2 | 13
  AE of Grade ≥ 4 | 0 | 2 | 6
  Serious adverse event (SAE) | 9 | 2 | 12
  Fatal adverse events | 0 | 0 | 2
  Led to discontinuation of study drug | 3 | 1 | 2
  Led to interruption of study drug | 4 | 1 | 6
  Related adverse events | 9 | 2 | 11
  Related AE Grade ≥ 3 | 5 | 2 | 5
  Related AE Grade ≥ 4 | 0 | 1 | 2
  Serious related adverse events | 5 | 2 | 3
  Related AE led to discontinuation of study drug | 2 | 1 | 2
  Related AE led to interruption of study drug | 3 | 1 | 3

10. Secondary Outcome: Blinatumomab Steady State Serum Concentration
Description: Blinatumomab serum levels were analyzed using a validated cluster of differentiation (CD)69 activation bioassay with a lower limit of quantification (LLOQ) of 50 pg/mL. Steady-state concentration (Css) was based on actual dose received, rather than based on cohort or time or day.
Time Frame: Cycle 1: predose; Day 3 and Day 8 (Css for 9 ug/day); Day 15 (Css for 28 ug/day); and Day 29, Day 43 and Day 57 (Css for 112 ug/day)
Population: Pharmacokinetic (PK) data set (all participants who received any infusion of blinatumomab and had at least one PK sample collected).
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Blinatumomab 9 μg/d: Participants received blinatumomab administered via a continuous intravenous infusion (CIV) 9 µg/day.
- Blinatumomab 28 μg/d: Participants received blinatumomab CIV 28 µg/day.
- Blinatumomab 112 μg/d: Participants received blinatumomab administered CIV 112 µg/day.
Arm/Group | Blinatumomab 9 μg/d | Blinatumomab 28 μg/d | Blinatumomab 112 μg/d
Number analyzed (Participants) | 20 | 16 | 12
pg/mL | 277 (210) | 565 (208) | 2800 (1150)

11. Secondary Outcome: Leukocyte Counts
Description: Leukocyte (white blood cells) counts were analyzed by differential blood count analysis.
Time Frame: Screening (Day -20 to Day 0), Day 1 pre-infusion, Days 8, 15, 29, 43, end of infusion (day 53), end of core study (day 87), and follow-up at 3, 6, 9, 12, 15, 18, 21 and 24 months after the first response assessment
Population: Enrolled participants with available data at each time point. All participants are included in pre-infusion and follow-up data points, only those participants in Cohorts 1 and 3 who had the same treatment schedule of 9/28/112 µg/day step dosing are included in the infusion time points (day 8 through end of infusion).
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Groups:
- Blinatumomab: All participants who received blinatumomab by continuous intravenous infusion during the core study.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 6.376 (3.284)
  Day 1 Prior (N = 24) | 5.729 (2.891)
  Day 8 (N = 21) | 6.819 (3.201)
  Day 15 (N = 16) | 6.400 (2.486)
  Day 29 (N = 11) | 3.764 (2.160)
  Day 43 (N = 8) | 4.950 (3.819)
  End of Infusion (N = 9) | 4.611 (2.114)
  End of Core Study (N = 6) | 6.850 (2.818)
  3-Month Follow-up (N = 5) | 4.820 (1.616)
  6-Month Follow-up (N = 6) | 5.183 (1.380)
  9-Month Follow-up (N = 4) | 4.425 (0.854)
  12-Month Follow-up (N = 4) | 5.700 (1.424)
  15-Month Follow-up (N = 3) | 4.767 (0.874)
  18-Month Follow-up (N = 3) | 6.467 (1.779)
  21-Month Follow-up (N = 21) | 5.450 (0.495)
  24-Month Follow-up (N = 3) | 4.533 (1.069)

12. Secondary Outcome: Lymphocyte Counts
Description: Lymphocyte counts were analyzed by differential blood count analysis.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.779 (0.425)
  Day 1 Prior (N = 24) | 0.491 (0.259)
  Day 8 (N = 21) | 0.382 (0.215)
  Day 15 (N = 16) | 0.277 (0.165)
  Day 29 (N = 11) | 0.472 (0.273)
  Day 43 (N = 8) | 0.847 (0.511)
  End of Infusion (N = 9) | 0.767 (0.505)
  End of Core Study (N = 6) | 1.060 (0.489)
  3-Month Follow-up (N = 5) | 1.053 (0.421)
  6-Month Follow-up (N = 6) | 1.120 (0.621)
  9-Month Follow-up (N = 4) | 1.048 (0.381)
  12-Month Follow-up (N = 4) | 1.120 (0.449)
  15-Month Follow-up (N = 3) | 0.998 (0.527)
  18-Month Follow-up (N = 3) | 0.565 (0.180)
  21-Month Follow-up (N = 21) | 1.205 (0.839)
  24-Month Follow-up (N = 3) | 0.737 (0.478)

13. Secondary Outcome: Monocyte Counts
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.638 (0.415)
  Day 1 Prior (N = 24) | 0.300 (0.565)
  Day 8 (N = 21) | 0.202 (0.386)
  Day 15 (N = 16) | 0.188 (0.317)
  Day 29 (N = 11) | 0.318 (0.185)
  Day 43 (N = 8) | 0.646 (0.375)
  End of Infusion (N = 9) | 0.473 (0.241)
  End of Core Study (N = 6) | 0.711 (0.569)
  3-Month Follow-up (N = 5) | 0.585 (0.280)
  6-Month Follow-up (N = 6) | 0.487 (0.239)
  9-Month Follow-up (N = 4) | 0.452 (0.112)
  12-Month Follow-up (N = 4) | 0.469 (0.061)
  15-Month Follow-up (N = 3) | 0.511 (0.053)
  18-Month Follow-up (N = 3) | 0.290 (0.123)
  21-Month Follow-up (N = 21) | 0.516 (0.008)
  24-Month Follow-up (N = 3) | 0.234 (0.176)

14. Secondary Outcome: Granulocyte Count
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 4.968 (3.187)
  Day 1 Prior (N = 24) | 4.910 (2.425)
  Day 8 (N = 21) | 6.235 (2.881)
  Day 15 (N = 16) | 5.935 (2.387)
  Day 29 (N = 11) | 2.974 (2.019)
  Day 43 (N = 8) | 3.457 (3.395)
  End of Infusion (N = 9) | 3.353 (2.134)
  End of Core Study (N = 6) | 5.080 (3.012)
  3-Month Follow-up (N = 5) | 3.182 (1.117)
  6-Month Follow-up (N = 6) | 3.594 (0.950)
  9-Month Follow-up (N = 4) | 2.925 (0.675)
  12-Month Follow-up (N = 4) | 4.111 (1.382)
  15-Month Follow-up (N = 3) | 3.258 (0.745)
  18-Month Follow-up (N = 3) | 5.612 (1.713)
  21-Month Follow-up (N = 21) | 3.729 (0.352)
  24-Month Follow-up (N = 3) | 3.563 (0.711)

15. Secondary Outcome: CD19+ B-Cell Count
Description: CD19+ B-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.026 (0.072)
  Day 1 Prior (N = 24) | 0.029 (0.085)
  Day 8 (N = 21) | 0.001 (0.002)
  Day 15 (N = 16) | 0.000 (0.001)
  Day 29 (N = 11) | 0.000 (0.000)
  Day 43 (N = 8) | 0.000 (0.001)
  End of Infusion (N = 9) | 0.001 (0.001)
  End of Core Study (N = 6) | 0.001 (0.002)
  3-Month Follow-up (N = 5) | 0.025 (0.026)
  6-Month Follow-up (N = 6) | 0.029 (0.043)
  9-Month Follow-up (N = 4) | 0.054 (0.066)
  12-Month Follow-up (N = 4) | 0.082 (0.113)
  15-Month Follow-up (N = 3) | 0.094 (0.118)
  18-Month Follow-up (N = 3) | 0.071 (0.075)
  21-Month Follow-up (N = 21) | 0.131 (0.170)
  24-Month Follow-up (N = 3) | 0.108 (0.120)

16. Secondary Outcome: CD19+ B-Cells as a Percentage of All Lymphocytes
Description: CD19+ B-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of lymphocytes
  Screening (N = 25) | 2 (7)
  Day 1 Prior (N = 24) | 4 (9)
  Day 8 (N = 21) | 0 (0)
  Day 15 (N = 16) | 0 (0)
  Day 29 (N = 11) | 0 (0)
  Day 43 (N = 8) | 0 (0)
  End of Infusion (N = 9) | 0 (0)
  End of Core Study (N = 6) | 0 (0)
  3-Month Follow-up (N = 5) | 2 (2)
  6-Month Follow-up (N = 6) | 2 (3)
  9-Month Follow-up (N = 4) | 5 (5)
  12-Month Follow-up (N = 4) | 7 (9)
  15-Month Follow-up (N = 3) | 7 (7)
  18-Month Follow-up (N = 3) | 11 (9)
  21-Month Follow-up (N = 21) | 8 (8)
  24-Month Follow-up (N = 3) | 12 (7)

17. Secondary Outcome: CD3+ T-Cell Count
Description: CD3+ T-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.578 (0.355)
  Day 1 Prior (N = 24) | 0.349 (0.233)
  Day 8 (N = 21) | 0.282 (0.194)
  Day 15 (N = 16) | 0.199 (0.159)
  Day 29 (N = 11) | 0.348 (0.231)
  Day 43 (N = 8) | 0.613 (0.426)
  End of Infusion (N = 9) | 0.543 (0.421)
  End of Core Study (N = 6) | 0.825 (0.431)
  3-Month Follow-up (N = 5) | 0.773 (0.443)
  6-Month Follow-up (N = 6) | 0.782 (0.345)
  9-Month Follow-up (N = 4) | 0.671 (0.184)
  12-Month Follow-up (N = 4) | 0.703 (0.203)
  15-Month Follow-up (N = 3) | 0.594 (0.227)
  18-Month Follow-up (N = 3) | 0.298 (0.049)
  21-Month Follow-up (N = 21) | 0.623 (0.266)
  24-Month Follow-up (N = 3) | 0.456 (0.257)

18. Secondary Outcome: CD3+ T-Cells as a Percentage of All Lymphocytes
Description: CD3+ T-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of lymphocytes
  Screening (N = 25) | 72 (14)
  Day 1 Prior (N = 24) | 68 (18)
  Day 8 (N = 21) | 70 (19)
  Day 15 (N = 16) | 67 (19)
  Day 29 (N = 11) | 73 (15)
  Day 43 (N = 8) | 71 (13)
  End of Infusion (N = 9) | 66 (14)
  End of Core Study (N = 6) | 76 (16)
  3-Month Follow-up (N = 5) | 73 (11)
  6-Month Follow-up (N = 6) | 66 (21)
  9-Month Follow-up (N = 4) | 66 (6)
  12-Month Follow-up (N = 4) | 65 (9)
  15-Month Follow-up (N = 3) | 61 (7)
  18-Month Follow-up (N = 3) | 57 (20)
  21-Month Follow-up (N = 21) | 58 (16)
  24-Month Follow-up (N = 3) | 63 (8)

19. Secondary Outcome: CD4+ T-Cell Count
Description: CD4+ T-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.254 (0.160)
  Day 1 Prior (N = 24) | 0.152 (0.128)
  Day 8 (N = 21) | 0.131 (0.128)
  Day 15 (N = 16) | 0.085 (0.084)
  Day 29 (N = 11) | 0.170 (0.172)
  Day 43 (N = 8) | 0.261 (0.219)
  End of Infusion (N = 9) | 0.241 (0.254)
  End of Core Study (N = 6) | 0.375 (0.251)
  3-Month Follow-up (N = 5) | 0.371 (0.216)
  6-Month Follow-up (N = 6) | 0.371 (0.237)
  9-Month Follow-up (N = 4) | 0.309 (0.184)
  12-Month Follow-up (N = 4) | 0.399 (0.193)
  15-Month Follow-up (N = 3) | 0.326 (0.220)
  18-Month Follow-up (N = 3) | 0.178 (0.042)
  21-Month Follow-up (N = 21) | 0.373 (0.279)
  24-Month Follow-up (N = 3) | 0.258 (0.248)

20. Secondary Outcome: CD4+ T-Cells as a Percentage of All Lymphocytes
Description: CD4+ T-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of lymphocytes
  Screening (N = 25) | 33 (11)
  Day 1 Prior (N = 24) | 28 (14)
  Day 8 (N = 21) | 32 (17)
  Day 15 (N = 16) | 29 (13)
  Day 29 (N = 11) | 34 (18)
  Day 43 (N = 8) | 30 (12)
  End of Infusion (N = 9) | 28 (13)
  End of Core Study (N = 6) | 32 (15)
  3-Month Follow-up (N = 5) | 33 (9)
  6-Month Follow-up (N = 6) | 30 (10)
  9-Month Follow-up (N = 4) | 31 (13)
  12-Month Follow-up (N = 4) | 35 (7)
  15-Month Follow-up (N = 3) | 31 (7)
  18-Month Follow-up (N = 3) | 32 (6)
  21-Month Follow-up (N = 21) | 29 (4)
  24-Month Follow-up (N = 3) | 34 (8)

21. Secondary Outcome: CD8+ T-Cell Count
Description: CD8+ T-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.298 (0.256)
  Day 1 Prior (N = 24) | 0.186 (0.136)
  Day 8 (N = 21) | 0.134 (0.099)
  Day 15 (N = 16) | 0.102 (0.095)
  Day 29 (N = 11) | 0.140 (0.076)
  Day 43 (N = 8) | 0.299 (0.237)
  End of Infusion (N = 9) | 0.284 (0.195)
  End of Core Study (N = 6) | 0.438 (0.284)
  3-Month Follow-up (N = 5) | 0.381 (0.254)
  6-Month Follow-up (N = 6) | 0.403 (0.304)
  9-Month Follow-up (N = 4) | 0.225 (0.039)
  12-Month Follow-up (N = 4) | 0.310 (0.200)
  15-Month Follow-up (N = 3) | 0.214 (0.023)
  18-Month Follow-up (N = 3) | 0.105 (0.057)
  21-Month Follow-up (N = 21) | 0.185 (0.026)
  24-Month Follow-up (N = 3) | 0.187 (0.068)

22. Secondary Outcome: CD8+ T-Cells as a Percentage of All Lymphocytes
Description: CD8+ T-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of lymphocytes
  Screening (N = 25) | 37 (18)
  Day 1 Prior (N = 24) | 37 (19)
  Day 8 (N = 21) | 35 (19)
  Day 15 (N = 16) | 35 (17)
  Day 29 (N = 11) | 33 (17)
  Day 43 (N = 8) | 37 (15)
  End of Infusion (N = 9) | 36 (16)
  End of Core Study (N = 6) | 43 (23)
  3-Month Follow-up (N = 5) | 36 (19)
  6-Month Follow-up (N = 6) | 34 (16)
  9-Month Follow-up (N = 4) | 25 (11)
  12-Month Follow-up (N = 4) | 28 (13)
  15-Month Follow-up (N = 3) | 24 (9)
  18-Month Follow-up (N = 3) | 21 (13)
  21-Month Follow-up (N = 21) | 20 (12)
  24-Month Follow-up (N = 3) | 27 (16)

23. Secondary Outcome: CD19+ B-Cell to CD3+ T-Cell Ratio
Description: CD19+ B-cells and CD3+ T-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
ratio
  Screening (N = 25) | 0.04 (0.15)
  Day 1 Prior (N = 24) | 0.07 (0.24)
  Day 8 (N = 21) | 0.00 (0.01)
  Day 15 (N = 16) | 0.00 (0.00)
  Day 29 (N = 11) | 0.00 (0.00)
  Day 43 (N = 8) | 0.00 (0.00)
  End of Infusion (N = 9) | 0.00 (0.01)
  End of Core Study (N = 6) | 0.00 (0.00)
  3-Month Follow-up (N = 5) | 0.03 (0.03)
  6-Month Follow-up (N = 6) | 0.04 (0.05)
  9-Month Follow-up (N = 4) | 0.08 (0.08)
  12-Month Follow-up (N = 4) | 0.12 (0.15)
  15-Month Follow-up (N = 3) | 0.13 (0.13)
  18-Month Follow-up (N = 3) | 0.25 (0.30)
  21-Month Follow-up (N = 21) | 0.17 (0.20)
  24-Month Follow-up (N = 3) | 0.19 (0.13)

24. Secondary Outcome: CD4+ T-Cell to CD8+ T-Cell Ratio
Description: CD4+ T-cells and CD8+ T-cell counts were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
ratio
  Screening (N = 25) | 1.32 (1.19)
  Day 1 Prior (N = 24) | 1.16 (1.45)
  Day 8 (N = 21) | 1.20 (0.96)
  Day 15 (N = 16) | 1.03 (0.71)
  Day 29 (N = 11) | 1.43 (1.08)
  Day 43 (N = 8) | 0.96 (0.53)
  End of Infusion (N = 9) | 1.09 (1.00)
  End of Core Study (N = 6) | 1.03 (0.80)
  3-Month Follow-up (N = 5) | 1.18 (0.79)
  6-Month Follow-up (N = 6) | 1.10 (0.70)
  9-Month Follow-up (N = 4) | 1.53 (1.25)
  12-Month Follow-up (N = 4) | 1.70 (1.47)
  15-Month Follow-up (N = 3) | 1.47 (0.81)
  18-Month Follow-up (N = 3) | 2.23 (1.70)
  21-Month Follow-up (N = 21) | 1.85 (1.34)
  24-Month Follow-up (N = 3) | 1.73 (1.21)

25. Secondary Outcome: CD4+ Naive T Cell Count
Description: CD4+ naive T-cell counts are native T-cells characterized by the cell-surface expression of CD197 and CD45RA and were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.028 (0.056)
  Day 1 Prior (N = 24) | 0.013 (0.022)
  Day 8 (N = 21) | 0.014 (0.033)
  Day 15 (N = 16) | 0.012 (0.024)
  Day 29 (N = 11) | 0.032 (0.071)
  Day 43 (N = 8) | 0.036 (0.060)
  End of Infusion (N = 9) | 0.037 (0.088)
  End of Core Study (N = 6) | 0.050 (0.083)
  3-Month Follow-up (N = 5) | 0.015 (0.019)
  6-Month Follow-up (N = 6) | 0.023 (0.044)
  9-Month Follow-up (N = 4) | 0.053 (0.090)
  12-Month Follow-up (N = 4) | 0.053 (0.084)
  15-Month Follow-up (N = 3) | 0.044 (0.059)
  18-Month Follow-up (N = 3) | 0.035 (0.041)
  21-Month Follow-up (N = 21) | 0.098 (0.103)
  24-Month Follow-up (N = 3) | 0.016 (0.013)

26. Secondary Outcome: CD4+ Naive T Cells as a Percentage of All CD4+ T-Cells
Description: as for outcome 25
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD4+ T-cells
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of CD4+ T-cells
  Screening (N = 25) | 8 (9)
  Day 1 Prior (N = 24) | 7 (7)
  Day 8 (N = 21) | 7 (7)
  Day 15 (N = 16) | 10 (9)
  Day 29 (N = 11) | 9 (11)
  Day 43 (N = 8) | 10 (10)
  End of Infusion (N = 9) | 8 (9)
  End of Core Study (N = 6) | 9 (13)
  3-Month Follow-up (N = 5) | 4 (3)
  6-Month Follow-up (N = 6) | 4 (7)
  9-Month Follow-up (N = 4) | 11 (15)
  12-Month Follow-up (N = 4) | 12 (14)
  15-Month Follow-up (N = 3) | 10 (9)
  18-Month Follow-up (N = 3) | 19 (19)
  21-Month Follow-up (N = 21) | 23 (9)
  24-Month Follow-up (N = 3) | 8 (10)

27. Secondary Outcome: CD4+ Central Memory T-Cell (TCM) Count
Description: Central memory T cells are characterized by the cell-surface expression of CD197 but not CD45RA and were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.048 (0.053)
  Day 1 Prior (N = 24) | 0.029 (0.034)
  Day 8 (N = 21) | 0.027 (0.042)
  Day 15 (N = 16) | 0.014 (0.025)
  Day 29 (N = 11) | 0.032 (0.065)
  Day 43 (N = 8) | 0.032 (0.035)
  End of Infusion (N = 9) | 0.049 (0.103)
  End of Core Study (N = 6) | 0.062 (0.075)
  3-Month Follow-up (N = 5) | 0.019 (0.009)
  6-Month Follow-up (N = 6) | 0.027 (0.020)
  9-Month Follow-up (N = 4) | 0.043 (0.056)
  12-Month Follow-up (N = 4) | 0.065 (0.073)
  15-Month Follow-up (N = 3) | 0.039 (0.020)
  18-Month Follow-up (N = 3) | 0.033 (0.031)
  21-Month Follow-up (N = 21) | 0.056 (0.054)
  24-Month Follow-up (N = 3) | 0.021 (0.010)

28. Secondary Outcome: CD4+ TCM Cells as a Percentage of All CD4+ T-Cells
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD4+ T-cells
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of CD4+ T-cells
  Screening (N = 25) | 18 (12)
  Day 1 Prior (N = 24) | 20 (15)
  Day 8 (N = 21) | 19 (15)
  Day 15 (N = 16) | 14 (12)
  Day 29 (N = 11) | 13 (10)
  Day 43 (N = 8) | 13 (9)
  End of Infusion (N = 9) | 15 (11)
  End of Core Study (N = 6) | 14 (11)
  3-Month Follow-up (N = 5) | 6 (3)
  6-Month Follow-up (N = 6) | 9 (4)
  9-Month Follow-up (N = 4) | 11 (9)
  12-Month Follow-up (N = 4) | 18 (16)
  15-Month Follow-up (N = 3) | 13 (6)
  18-Month Follow-up (N = 3) | 18 (14)
  21-Month Follow-up (N = 21) | 14 (4)
  24-Month Follow-up (N = 3) | 12 (11)

29. Secondary Outcome: CD4+ Effector Memory T-Cell (TEM) Count
Description: Effector memory T cells are characterized by the lack of expression of CD197 and CD45RA and were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.161 (0.089)
  Day 1 Prior (N = 24) | 0.099 (0.096)
  Day 8 (N = 21) | 0.083 (0.076)
  Day 15 (N = 16) | 0.051 (0.044)
  Day 29 (N = 11) | 0.097 (0.059)
  Day 43 (N = 8) | 0.169 (0.117)
  End of Infusion (N = 9) | 0.140 (0.091)
  End of Core Study (N = 6) | 0.220 (0.142)
  3-Month Follow-up (N = 5) | 0.279 (0.153)
  6-Month Follow-up (N = 6) | 0.267 (0.158)
  9-Month Follow-up (N = 4) | 0.191 (0.037)
  12-Month Follow-up (N = 4) | 0.226 (0.100)
  15-Month Follow-up (N = 3) | 0.199 (0.087)
  18-Month Follow-up (N = 3) | 0.106 (0.066)
  21-Month Follow-up (N = 21) | 0.181 (0.107)
  24-Month Follow-up (N = 3) | 0.175 (0.133)

30. Secondary Outcome: CD4+ TEM Cells as a Percentage of All CD4+ T-Cells
Description: as for outcome 29
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD4+ T-cells
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of CD4+ T-cells
  Screening (N = 25) | 41 (19)
  Day 1 Prior (N = 24) | 39 (19)
  Day 8 (N = 21) | 36 (19)
  Day 15 (N = 16) | 46 (17)
  Day 29 (N = 11) | 34 (20)
  Day 43 (N = 8) | 39 (26)
  End of Infusion (N = 9) | 41 (24)
  End of Core Study (N = 6) | 41 (24)
  3-Month Follow-up (N = 5) | 46 (26)
  6-Month Follow-up (N = 6) | 41 (21)
  9-Month Follow-up (N = 4) | 42 (18)
  12-Month Follow-up (N = 4) | 40 (15)
  15-Month Follow-up (N = 3) | 46 (17)
  18-Month Follow-up (N = 3) | 43 (12)
  21-Month Follow-up (N = 21) | 45 (3)
  24-Month Follow-up (N = 3) | 51 (22)

31. Secondary Outcome: CD8+ Naive T-Cell Count
Description: CD8+ naive T-cell counts are native T-cells characterized by the cell-surface expression of CD197 and CD45RA and were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.029 (0.043)
  Day 1 Prior (N = 24) | 0.024 (0.050)
  Day 8 (N = 21) | 0.010 (0.012)
  Day 15 (N = 16) | 0.006 (0.005)
  Day 29 (N = 11) | 0.012 (0.014)
  Day 43 (N = 8) | 0.019 (0.036)
  End of Infusion (N = 9) | 0.011 (0.015)
  End of Core Study (N = 6) | 0.023 (0.018)
  3-Month Follow-up (N = 5) | 0.011 (0.007)
  6-Month Follow-up (N = 6) | 0.020 (0.022)
  9-Month Follow-up (N = 4) | 0.011 (0.012)
  12-Month Follow-up (N = 4) | 0.011 (0.009)
  15-Month Follow-up (N = 3) | 0.014 (0.011)
  18-Month Follow-up (N = 3) | 0.007 (0.008)
  21-Month Follow-up (N = 21) | 0.015 (0.006)
  24-Month Follow-up (N = 3) | 0.010 (0.009)

32. Secondary Outcome: CD8+ Naive T-Cells as a Percentage of All CD8+ T-Cells
Description: as for outcome 31
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD8+ T-cells
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of CD8+ T-cells
  Screening (N = 25) | 10 (10)
  Day 1 Prior (N = 24) | 12 (13)
  Day 8 (N = 21) | 9 (8)
  Day 15 (N = 16) | 8 (7)
  Day 29 (N = 11) | 8 (7)
  Day 43 (N = 8) | 6 (7)
  End of Infusion (N = 9) | 3 (3)
  End of Core Study (N = 6) | 6 (6)
  3-Month Follow-up (N = 5) | 4 (4)
  6-Month Follow-up (N = 6) | 5 (5)
  9-Month Follow-up (N = 4) | 6 (7)
  12-Month Follow-up (N = 4) | 6 (6)
  15-Month Follow-up (N = 3) | 6 (5)
  18-Month Follow-up (N = 3) | 10 (8)
  21-Month Follow-up (N = 21) | 8 (4)
  24-Month Follow-up (N = 3) | 10 (12)

33. Secondary Outcome: CD8+ TCM Cell Counts
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 100 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
100 cells/µL
  Screening (N = 25) | 0.020 (0.027)
  Day 1 Prior (N = 24) | 0.014 (0.021)
  Day 8 (N = 21) | 0.010 (0.013)
  Day 15 (N = 16) | 0.004 (0.005)
  Day 29 (N = 11) | 0.007 (0.007)
  Day 43 (N = 8) | 0.012 (0.015)
  End of Infusion (N = 9) | 0.009 (0.009)
  End of Core Study (N = 6) | 0.016 (0.023)
  3-Month Follow-up (N = 5) | 0.008 (0.003)
  6-Month Follow-up (N = 6) | 0.016 (0.014)
  9-Month Follow-up (N = 4) | 0.006 (0.004)
  12-Month Follow-up (N = 4) | 0.010 (0.010)
  15-Month Follow-up (N = 3) | 0.004 (0.002)
  18-Month Follow-up (N = 3) | 0.002 (0.001)
  21-Month Follow-up (N = 21) | 0.002 (0.001)
  24-Month Follow-up (N = 3) | 0.006 (0.004)

34. Secondary Outcome: CD8+ TCM Cells as a Percentage of All CD8+ T-Cells
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD8+ T-cells
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of CD8+ T-cells
  Screening (N = 25) | 7 (7)
  Day 1 Prior (N = 24) | 8 (11)
  Day 8 (N = 21) | 10 (13)
  Day 15 (N = 16) | 4 (5)
  Day 29 (N = 11) | 7 (10)
  Day 43 (N = 8) | 9 (18)
  End of Infusion (N = 9) | 5 (6)
  End of Core Study (N = 6) | 5 (8)
  3-Month Follow-up (N = 5) | 3 (2)
  6-Month Follow-up (N = 6) | 4 (3)
  9-Month Follow-up (N = 4) | 3 (2)
  12-Month Follow-up (N = 4) | 3 (3)
  15-Month Follow-up (N = 3) | 2 (1)
  18-Month Follow-up (N = 3) | 2 (1)
  21-Month Follow-up (N = 21) | 1 (0)
  24-Month Follow-up (N = 3) | 6 (8)

35. Secondary Outcome: CD8+ Effector Memory T-Cell (TEM) Count
Description: as for outcome 29
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.127 (0.162)
  Day 1 Prior (N = 24) | 0.075 (0.066)
  Day 8 (N = 21) | 0.065 (0.058)
  Day 15 (N = 16) | 0.045 (0.053)
  Day 29 (N = 11) | 0.067 (0.039)
  Day 43 (N = 8) | 0.135 (0.108)
  End of Infusion (N = 9) | 0.128 (0.077)
  End of Core Study (N = 6) | 0.180 (0.089)
  3-Month Follow-up (N = 5) | 0.146 (0.071)
  6-Month Follow-up (N = 6) | 0.179 (0.158)
  9-Month Follow-up (N = 4) | 0.116 (0.061)
  12-Month Follow-up (N = 4) | 0.174 (0.162)
  15-Month Follow-up (N = 3) | 0.095 (0.025)
  18-Month Follow-up (N = 3) | 0.049 (0.027)
  21-Month Follow-up (N = 21) | 0.085 (0.013)
  24-Month Follow-up (N = 3) | 0.054 (0.027)

36. Secondary Outcome: CD8+ TEM Cells as a Percentage of All CD8+ T-Cells
Description: as for outcome 29
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD8+ T-cells
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of CD8+ T-cells
  Screening (N = 25) | 42 (19)
  Day 1 Prior (N = 24) | 42 (17)
  Day 8 (N = 21) | 46 (18)
  Day 15 (N = 16) | 43 (13)
  Day 29 (N = 11) | 51 (19)
  Day 43 (N = 8) | 46 (23)
  End of Infusion (N = 9) | 51 (21)
  End of Core Study (N = 6) | 49 (22)
  3-Month Follow-up (N = 5) | 47 (23)
  6-Month Follow-up (N = 6) | 50 (24)
  9-Month Follow-up (N = 4) | 50 (21)
  12-Month Follow-up (N = 4) | 51 (13)
  15-Month Follow-up (N = 3) | 46 (15)
  18-Month Follow-up (N = 3) | 46 (7)
  21-Month Follow-up (N = 21) | 46 (1)
  24-Month Follow-up (N = 3) | 33 (9)

37. Secondary Outcome: CD8+ Terminally Differentiated Effector Memory T-cells (TEMRA) Count
Description: Terminally differentiated effector memory T cells are characterized by the cell-surface expression of CD45RA but not CD197 and were analyzed by flow cytometry.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 1000 cells/µL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
1000 cells/µL
  Screening (N = 25) | 0.123 (0.099)
  Day 1 Prior (N = 24) | 0.072 (0.069)
  Day 8 (N = 21) | 0.051 (0.042)
  Day 15 (N = 16) | 0.047 (0.048)
  Day 29 (N = 11) | 0.058 (0.050)
  Day 43 (N = 8) | 0.132 (0.126)
  End of Infusion (N = 9) | 0.135 (0.131)
  End of Core Study (N = 6) | 0.226 (0.249)
  3-Month Follow-up (N = 5) | 0.214 (0.220)
  6-Month Follow-up (N = 6) | 0.187 (0.182)
  9-Month Follow-up (N = 4) | 0.094 (0.046)
  12-Month Follow-up (N = 4) | 0.117 (0.065)
  15-Month Follow-up (N = 3) | 0.099 (0.041)
  18-Month Follow-up (N = 3) | 0.047 (0.035)
  21-Month Follow-up (N = 21) | 0.086 (0.016)
  24-Month Follow-up (N = 3) | 0.100 (0.084)

38. Secondary Outcome: CD8+ TEMRA Cells as a Percentage of All CD8+ T-Cells
Description: as for outcome 37
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of CD8+ T-cells
Arm/Group | Blinatumomab
Number analyzed (Participants) | 25
percentage of CD8+ T-cells
  Screening (N = 25) | 41 (19)
  Day 1 Prior (N = 24) | 39 (19)
  Day 8 (N = 21) | 36 (19)
  Day 15 (N = 16) | 46 (17)
  Day 29 (N = 11) | 34 (20)
  Day 43 (N = 8) | 39 (26)
  End of Infusion (N = 9) | 41 (24)
  End of Core Study (N = 6) | 41 (24)
  3-Month Follow-up (N = 5) | 46 (26)
  6-Month Follow-up (N = 6) | 41 (21)
  9-Month Follow-up (N = 4) | 42 (18)
  12-Month Follow-up (N = 4) | 40 (15)
  15-Month Follow-up (N = 3) | 46 (17)
  18-Month Follow-up (N = 3) | 43 (12)
  21-Month Follow-up (N = 21) | 45 (3)
  24-Month Follow-up (N = 3) | 51 (22)

ADVERSE EVENTS:
Time Frame: From the first dose of blinatumomab until up to 30 days after the last dose, until the data cut-off date of 10 July 2014; the overall median duration of treatment exposure was 46.8 days.
Description: Adverse Events were not pre-specified to be monitored/assessed after 10 July 2014.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Cohort 1: Blinatumomab 9/28/112 µg/d: Participants received blinatumomab administered CIV 9 µg/day for the first week, followed by 28 µg/day for the second week, then 112 µg/day for the remaining 6 weeks of treatment during Cycle 1. Participants who achieved a CR or PR, or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
- Cohort 2: Blinatumomab 112 µg/d: Participants received blinatumomab administered CIV at a constant dose of 112 µg/day for 8 weeks of treatment during Cycle 1. Participants who achieved CR or PR, or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
- Cohort 1+3: Blinatumomab 9/28/112µg/d: Participants received blinatumomab administered CIV 9 µg/day for the first week, followed by 28 µg/day for the second week, then 112 µg/day for the remaining 6 weeks of treatment during Cycle 1. Participants who achieved CR or PR, or had stable disease after the first treatment cycle were eligible to receive a second (consolidation) cycle of treatment over 4 weeks, following a 4-week treatment-free interval.
- Blinatumomab Overall: All participants who received blinatumomab by continuous intravenous infusion during the core study.
Arm/Group | Cohort 1: Blinatumomab 9/28/112 µg/d | Cohort 2: Blinatumomab 112 µg/d | Cohort 3: Blinatumomab 9/28/112 µg/d | Cohort 1+3: Blinatumomab 9/28/112µg/d | Blinatumomab Overall
Serious Adverse Events (participants affected / at risk) | 9/9 | 2/2 | 12/14 | 21/23 | 23/25
Other Adverse Events (participants affected / at risk) | 9/9 | 2/2 | 14/14 | 23/23 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Blinatumomab 9/28/112 µg/d (N=9) | Cohort 2: Blinatumomab 112 µg/d (N=2) | Cohort 3: Blinatumomab 9/28/112 µg/d (N=14) | Cohort 1+3: Blinatumomab 9/28/112µg/d (N=23) | Blinatumomab Overall (N=25)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 1 | 1
Pain (General disorders) | 1 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 2 | 3 | 4
Catheter site infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Device related infection (Infections and infestations) | 0 | 0 | 5 | 5 | 5
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 1 | 2 | 5 | 6
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Drug administration error (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Pancreatic enzymes increased (Investigations) | 0 | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Aphasia (Nervous system disorders) | 2 | 0 | 0 | 2 | 2
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 2 | 2
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 1 | 0 | 1 | 2
Speech disorder (Nervous system disorders) | 1 | 1 | 0 | 1 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Blinatumomab 9/28/112 µg/d (N=9) | Cohort 2: Blinatumomab 112 µg/d (N=2) | Cohort 3: Blinatumomab 9/28/112 µg/d (N=14) | Cohort 1+3: Blinatumomab 9/28/112µg/d (N=23) | Blinatumomab Overall (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 4 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 4 | 5 | 5
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 2 | 2
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 1 | 1
Keratitis (Eye disorders) | 1 | 0 | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 1 | 5 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 1
Catheter site erythema (General disorders) | 0 | 0 | 1 | 1 | 1
Catheter site rash (General disorders) | 0 | 0 | 1 | 1 | 1
Chills (General disorders) | 1 | 0 | 2 | 3 | 3
Disease progression (General disorders) | 0 | 0 | 3 | 3 | 3
Facial pain (General disorders) | 0 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 3 | 1 | 3 | 6 | 7
General physical health deterioration (General disorders) | 1 | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1 | 1
Oedema (General disorders) | 1 | 0 | 5 | 6 | 6
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 1
Pain (General disorders) | 0 | 0 | 1 | 1 | 1
Pyrexia (General disorders) | 4 | 1 | 5 | 9 | 10
Ulcer (General disorders) | 1 | 0 | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Candida infection (Infections and infestations) | 2 | 0 | 0 | 2 | 2
Candiduria (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Fungal infection (Infections and infestations) | 1 | 1 | 0 | 1 | 2
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 3 | 3
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1
Antithrombin III decreased (Investigations) | 0 | 0 | 1 | 1 | 1
Blood fibrinogen increased (Investigations) | 0 | 0 | 1 | 1 | 1
Blood glucose increased (Investigations) | 0 | 0 | 4 | 4 | 4
Blood immunoglobulin G decreased (Investigations) | 2 | 0 | 0 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 1 | 1
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 1 | 1
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 3 | 4 | 4
Corneal reflex decreased (Investigations) | 0 | 0 | 1 | 1 | 1
Fibrin D dimer increased (Investigations) | 1 | 0 | 1 | 2 | 2
Fibrinolysis increased (Investigations) | 1 | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 1
PO2 decreased (Investigations) | 1 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 3 | 3 | 3
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 4 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 4 | 4
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 2
Dyscalculia (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Hyporeflexia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 2 | 2
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 2 | 2
Speech disorder (Nervous system disorders) | 3 | 1 | 0 | 3 | 4
Tremor (Nervous system disorders) | 6 | 2 | 4 | 10 | 12
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 2 | 2
Disorientation (Psychiatric disorders) | 2 | 1 | 0 | 2 | 3
Encopresis (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1
Fear (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 2 | 2
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 2 | 2 | 2
Enuresis (Renal and urinary disorders) | 2 | 0 | 0 | 2 | 2
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 2 | 2
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 4 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Embolism (Vascular disorders) | 1 | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.